CLINICAL TRIAL: NCT01202773
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of LY2127399 in Patients With Moderate to Severe Rheumatoid Arthritis (RA) Who Had an Inadequate Response to One or More TNF-α Inhibitors (FLEX V)
Brief Title: A Study in Participants With Rheumatoid Arthritis
Acronym: FLEX V
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated not based on safety concerns, but due to insufficient efficacy.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13732; H9B-MC-BCDV (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-09-14; First posted 2010-09-16 (Estimated); Results first posted 2018-05-14 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tabalumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 120 milligrams (mg) LY2127399 (Experimental): Given every 4 weeks (Q4W) for 24 weeks. Participants receive a 240-mg loading dose when initiating treatment.
  During the Treatment Period, for blinding purposes, participants will alternate injections of LY2127399 and injections of placebo every 2 weeks (Q2W).
  At Week 16, responders will receive 1 injection of 120 mg of LY2127399 and 1 injection of placebo, followed by 120 mg of LY2127399 Q4W for the rest of the 24-week treatment period.
  At Week 16, non-responders (NR) will receive 1 injection of 90 mg of LY2127399 and 1 injection of placebo, followed by 90 mg of LY2127399 Q2W for the rest of the 24-week treatment period.
  Interventions: Drug: LY2127399; Drug: Placebo Q4W
- 90 mg LY2127399 (Experimental): Given Q2W for 24 weeks. Participants receive a 180-mg loading dose when initiating treatment.
  At Week 16, both responders and NR will receive 1 injection of 90 mg of LY2127399 and 1 injection of placebo, followed by 90 mg of LY2127399 Q2W for the rest of the 24-week treatment period.
  Interventions: Drug: LY2127399
- Placebo (Placebo Comparator): Given Q2W for 24 weeks. Participants receive 2 injections of placebo when initiating treatment.
  At Week 16, responders will receive 2 injections of placebo, followed by 1 injection of placebo Q2W for the rest of the 24-week treatment period.
  At Week 16, NR will receive a 180-mg loading dose of LY2127399 (2 injections of 90 mg), followed by 90 mg of LY2127399 Q2W for the rest of the 24-week treatment period.
  Interventions: Drug: LY2127399; Drug: Placebo Q2W

INTERVENTIONS:
Drug: LY2127399 — Administered Subcutaneously (SC)
Drug: Placebo Q4W — Administered SC
  Arms: 120 milligrams (mg) LY2127399
Drug: Placebo Q2W — Administered SC
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to help answer if LY2127399 is safe and effective in the treatment of rheumatoid arthritis in participants with an inadequate response to one or more tumor necrosis factor-alpha (TNF-α) inhibitors.

This study is comprised of 2 periods:

Period 1: 24-week blinded treatment

Period 2: 48-week post-treatment follow-up

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RA of more than 6 months and less than 15 years
* At least 8 tender and swollen joints
* An abnormally high C-reactive protein (CRP) level or erythrocyte sedimentation rate (ESR)
* Positive for rheumatoid factor (RF) or anti-cyclic citrullinated peptide (CCP) antibody
* Previously treated with biologic TNF-α inhibitor therapy (infliximab, certolizumab, golimumab, etanercept, adalimumab) and stopped treatment due to insufficient efficacy or intolerance
* Regular use of at least 1 conventional disease-modifying anti-rheumatic drug (DMARD), with a stable dose for at least 8 weeks prior to study start
* Woman must not be pregnant, breastfeeding, or become pregnant during the study

Exclusion Criteria:

* Use of unstable doses of non-steroidal anti-inflammatory drugs (NSAIDS) in the past 6 weeks
* Steroid injection or intravenous (IV) infusion in the last 6 weeks
* Use of more than 10 milligrams/day (mg/day) of oral steroids in the last 6 weeks
* History of a serious reaction to other biological DMARDs
* Use of an oral calcineurin inhibitor (for example, cyclosporin or tacrolimus) in the last 8 weeks
* Surgery on a joint or other major surgery less than 2 months ago, or plans to have joint surgery or major surgery during the study
* Active fibromyalgia, juvenile chronic arthritis, spondyloarthropathy, Crohn's disease, ulcerative colitis, psoriatic arthritis, or other systemic inflammatory condition except RA
* Cervical cancer or squamous skin cancer within the past 3 years, or other cancer within the past 5 years
* Received a live vaccine received within the past 12 weeks (for example, vaccines for measles, mumps, rubella, and chicken pox, and nasal-spray flu vaccines)
* Hepatitis or human immunodeficiency virus (HIV)
* A serious bacterial infection (for example, pneumonia or cellulitis) within 3 months or a serious bone or joint infection within 6 months
* Symptoms of herpes zoster or herpes simplex within the last month
* Active or latent tuberculosis (TB)
* Current symptoms of a serious disorder or illness
* Use of an investigational drug within the last month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456 (Actual)
Dates: Start 2011-01; Primary Completion 2013-03 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (201):
- United States (110):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Huntsville, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paradise Valley, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Phoenix, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Scottsdale, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jonesboro, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Little Rock, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Escondido, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fresno, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hemet, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Huntington Beach, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Mesa, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Loma Linda, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Long Beach, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Angeles, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Diego, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Monica, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Torrance, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tustin, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Upland, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Whittier, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wildomar, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Colorado Springs, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Denver, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lewes, Delaware
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aventura, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boca Raton, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boynton Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., DeBary, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Port Richey, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palm Harbor, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pinellas Park, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tamarac, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampa, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Venice, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vero Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Palm Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Decatur, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dunwoody, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gainesville, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marietta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stockbridge, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Eagle, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Idaho Falls, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Peoria, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rock Island, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brownsburg, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Evansville, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kansas City, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bowling Green, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lexington, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Owensboro, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monroe, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wheaton, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Haverhill, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Worcester, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Clair Shores, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edina, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Flowood, Mississippi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jackson, Mississippi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cape Girardeau, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Florissant, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kalispell, Montana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashua, New Hampshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berkeley Heights, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Clifton, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albuquerque, New Mexico
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brooklyn, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charlotte, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greensboro, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hickory, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sanford, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bismarck, North Dakota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cleveland, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tulsa, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bethlehem, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Erie, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Limerick, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wexford, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbia, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greenville, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greer, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Myrtle Beach, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taylors, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Knoxville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Austin, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lubbock, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mesquite, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sugar Land, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Burlington, Vermont
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chesapeake, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Danville, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Richmond, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spokane, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tacoma, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wenatchee, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Clarksburg, West Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milwaukee, Wisconsin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Racine, Wisconsin
- Argentina (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Córdoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Luján
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mar del Plata
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Quilmes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Isidro
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Miguel de Tucumán
- Australia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kogarah, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Herston, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Malvern East
- Brazil (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Campinas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Goiânia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Juiz de Fora
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., São Paulo
- Colombia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bogotá
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Medellín
- France (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montpellier
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orléans
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint-Etienne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Strasbourg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toulouse
- Germany (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bad Doberan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bad Nauheim
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baden-Baden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cologne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dresden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Erlangen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frankfurt
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Göttingen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Munich
- Greece (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Haidari/Athens
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heraklion
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Larissa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Thessaloniki
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arenzano, Italy
- Japan (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gunma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miyazaki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagasaki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Okayama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
- Malaysia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Perak
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Putrajaya
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sarawak
- Mexico (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chihuahua City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Col Centro
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Querétaro
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Luis Potosí City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tlalpan
- New Zealand (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamilton
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rotorua
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tauranga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Timaru
- Poland (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bydgoszcz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Elblag
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lublin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Płock
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Torun
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
- Russia (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kazan'
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Khanty-Mansiysk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kursk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nizhny Novgorod
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Petrozavodsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stavropol
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Voronezh
- South Africa (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Benoni
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bloemfontein
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Limpopo
- South Korea (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Incheon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Suwon
- Spain (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., A Coruña
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bilboa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Manises
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santiago de Compostela
- Taiwan (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Keelung
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taichung
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei

REFERENCES:
- [Derived] Schiff M, Combe B, Dorner T, Kremer JM, Huizinga TW, Veenhuizen M, Gill A, Komocsar W, Berclaz PY, Ortmann R, Lee C. Efficacy and safety of tabalumab, an anti-BAFF monoclonal antibody, in patients with moderate-to-severe rheumatoid arthritis and inadequate response to TNF inhibitors: results of a randomised, double-blind, placebo-controlled, phase 3 study. RMD Open. 2015 Aug 12;1(1):e000037. doi: 10.1136/rmdopen-2014-000037. eCollection 2015. PMID 26535134

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study had a treatment period (Weeks 0-24) and a post-treatment follow-up period (24-48 weeks in length). All participants were assessed for nonresponse at Week 16 with non-responders (NR) defined as participants with <20% improvement from baseline in both tender and swollen joint counts.
Groups:
- 120 mg LY2127399: A loading dose of 240 milligrams (mg) (2 injections of 120 mg) of LY2127399 followed by maintenance dosing of 120 mg of LY2127399 administered subcutaneously (SC) every 4 weeks (Q4W) for 24 weeks. At Week 16, responders received 1 injection of 120 mg of LY2127399 and 1 injection of placebo, followed by 120 mg of LY2127399 Q4W for the rest of the 24-week treatment period. For blinding purposes, participants alternated injections of LY2127399 and injections of placebo every 2 weeks (Q2W).
  At Week 16, NR received 1 injection of 90 mg of LY2127399 and 1 injection of placebo, followed by 90 mg of LY2127399 Q2W for the rest of the 24-week treatment period.
- 90 mg LY2127399: A loading dose of 180 mg of LY2127399 (2 injections of 90 mg) followed by maintenance dosing of 90 mg of LY2127399 administered SC Q2W for 24 weeks.
  At Week 16, both responders and NR received 1 injection of 90 mg of LY2127399 and 1 injection of placebo, followed by 90 mg of LY2127399 Q2W for the rest of the 24-week treatment period.
- Placebo: A loading dose of 2 injections of placebo followed by maintenance dosing of 1 injection of placebo administered SC Q2W for 24 weeks. At Week 16, responders received 2 injections of placebo, followed by 1 injection of placebo Q2W for the rest of the 24-week treatment period.
  At Week 16, NR received a loading dose of 180 mg of LY2127399 (2 injections of 90 mg), followed by 90 mg of LY2127399 Q2W for the rest of the 24-week treatment period.
Period: Overall Study
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Started | 153 | 148 | 155
Received at Least 1 Dose of Study Drug | 153 | 147 | 154
Week 16 NR | 23 | 33 | 37
Post-Treatment Follow-Up Population | 46 | 36 | 51
Completed | 96 (Those who completed 24-week treatment period including both Week 16 responders and NR.) | 105 (Those who completed 24-week treatment period including both Week 16 responders and NR.) | 100 (Those who completed 24-week treatment period including both Week 16 responders and NR.)
Not Completed | 57 | 43 | 55
Not completed — Adverse Event | 4 | 5 | 5
Not completed — Lack of Efficacy | 5 | 4 | 9
Not completed — Entry Criteria Not Met | 2 | 0 | 1
Not completed — Lost to Follow-up | 1 | 2 | 2
Not completed — Withdrawal by Subject | 13 | 6 | 5
Not completed — Physician Decision | 2 | 0 | 0
Not completed — Protocol Violation | 11 | 6 | 10
Not completed — Sponsor Decision | 19 | 20 | 23

BASELINE CHARACTERISTICS:
Population: All randomized participants, including participants who did not take the assigned treatment, did not receive the correct treatment, or otherwise did not follow the protocol.
Groups:
- 120 mg LY2127399: A loading dose of 240 mg (2 injections of 120 mg) of LY2127399 followed by maintenance dosing of 120 mg of LY2127399 administered SC Q4W for 24 weeks. At Week 16, responders received 1 injection of 120 mg of LY2127399 and 1 injection of placebo, followed by 120 mg of LY2127399 Q4W for the rest of the 24-week treatment period. For blinding purposes, participants alternated injections of LY2127399 and injections of placebo Q2W.
  At Week 16, NR received 1 injection of 90 mg of LY2127399 and 1 injection of placebo, followed by 90 mg of LY2127399 Q2W for the rest of the 24-week treatment period.
- Total: Total of all reporting groups
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo | Total
Number analyzed (Participants) | 153 | 148 | 155 | 456
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (11.6) | 51.3 (11.7) | 54.0 (11.1) | 53.2 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 126 | 131 | 381
  Male | 29 | 22 | 24 | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 39 | 36 | 33 | 108
  Not Hispanic or Latino | 93 | 95 | 101 | 289
  Unknown or Not Reported | 21 | 17 | 21 | 59
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 8 | 9 | 6 | 23
  Asian | 10 | 9 | 13 | 32
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 14 | 16 | 18 | 48
  White | 119 | 108 | 112 | 339
  More than one race | 0 | 4 | 2 | 6
  Unknown or Not Reported | 2 | 2 | 4 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 89 | 90 | 89 | 268
  Taiwan | 0 | 0 | 1 | 1
  Greece | 2 | 1 | 1 | 4
  Spain | 2 | 2 | 2 | 6
  Russia | 6 | 4 | 4 | 14
  Colombia | 10 | 7 | 12 | 29
  France | 1 | 1 | 1 | 3
  Mexico | 3 | 3 | 2 | 8
  Argentina | 5 | 4 | 4 | 13
  Malaysia | 0 | 0 | 1 | 1
  Brazil | 7 | 7 | 7 | 21
  Poland | 14 | 14 | 14 | 42
  Australia | 0 | 1 | 2 | 3
  South Africa | 0 | 0 | 1 | 1
  Germany | 3 | 4 | 3 | 10
  New Zealand | 2 | 2 | 1 | 5
  Japan | 6 | 6 | 6 | 18
  South Korea | 3 | 2 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With American College of Rheumatology 20% (ACR20) Response
Description: ACR Responder Index: composite of clinical, laboratory, and functional measures of rheumatoid arthritis (RA). ACR20 Responder: a ≥20% improvement from baseline in both 68 tender joint counts (TJC) and 66 swollen joint counts (SJC) and a ≥20% improvement in at least 3 of 5 criteria: participant's and physician's global assessment of disease activity, Health Assessment Questionnaire-Disability Index (HAQ-DI) (which measured participants' perceived degree of difficulty performing daily activities), joint pain, and C-reactive protein (CRP). Percentage of participants achieving ACR20 response = (number of ACR20 responders / number of participants treated) * 100. All NR at Week 16, as well as all participants who discontinued study treatment at any time for any reason, were defined as NR starting at that time-point and going forward, including Week 24 endpoint.
Time Frame: Baseline through Week 24
Population: All randomized participants with evaluable ACR20 responder data. If participant's CRP was missing, last post-baseline value was used. If ACR was missing after carrying forward CRP, last post-baseline ACR response was used. Data after Week 16 for Week 16 NR were not included.
Measure: Number; unit: percentage of participants
Groups:
- 120 mg LY2127399: A loading dose of 240 mg (2 injections of 120 mg) of LY2127399 followed by maintenance dosing of 120 mg of LY2127399 administered SC Q4W for 24 weeks. At Week 16, responders received 1 injection of 120 mg of LY2127399 and 1 injection of placebo, followed by 120 mg of LY2127399 Q4W for the rest of the 24-week treatment period. For blinding purposes, participants alternated injections of LY2127399 and injections of placebo Q2W.
- 90 mg LY2127399: A loading dose of 180 mg of LY2127399 (2 injections of 90 mg) followed by maintenance dosing of 90 mg of LY2127399 administered SC Q2W for 24 weeks. At Week 16, responders received 1 injection of 90 mg of LY2127399 and 1 injection of placebo, followed by 90 mg of LY2127399 Q2W for the rest of the 24-week treatment period.
- Placebo: A loading dose of 2 injections of placebo followed by maintenance dosing of 1 injection of placebo administered SC Q2W for 24 weeks. At Week 16, responders received 2 injections of placebo, followed by 1 injection of placebo Q2W for the rest of the 24-week treatment period.
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 153 | 148 | 155
percentage of participants | 17.6 | 24.3 | 20.0

2. Secondary Outcome: Percentage of Participants With American College of Rheumatology 50% (ACR50) and 70% (ACR70) Response
Description: ACR Responder Index: composite of clinical, laboratory, and functional measures of RA. ACR50 Responder: had a ≥50% improvement from baseline in both 68 TJC and 66 SJC and a ≥50% improvement in at least 3 of 5 criteria: participant's (Pt's) and physician's global assessment of disease activity, HAQ-DI (measured Pts' perceived degree of difficulty performing daily activities), joint pain, and CRP. Percentage of Pt achieving ACR50 response = [number (No.) of ACR50 responders / No. of Pts treated]*100. ACR70 Responder: had a ≥70% improvement from baseline in both TJC and SJC and a ≥70% improvement in at least 3 of same 5 criteria for ACR50. Percentage of Pts achieving ACR70 response = (No. of ACR70 responders / No. of Pts treated)*100. All NR at Week 16, as well as all Pts who discontinued study treatment at any time for any reason, were defined as NR starting at that time-point and going forward, including Week 24 endpoint.
Time Frame: Baseline through Week 24
Population: All randomized participants with evaluable ACR50 or ACR70 responder data. If participant's CRP was missing, last post-baseline value was used. If ACR was missing after carrying forward CRP, last post-baseline ACR response was used. Data after Week 16 for Week 16 NR were not included.
Measure: Number; unit: percentage of participants
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 153 | 148 | 155
percentage of participants
  ACR50 | 7.2 | 5.4 | 3.9
  ACR70 | 2.6 | 2.0 | 0.6

3. Secondary Outcome: American College of Rheumatology Percent Improvement (ACR-N)
Description: ACR-N is a continuous measure of clinical, laboratory, and functional outcomes in RA that characterizes percentage (%) of improvement in disease activity from baseline based on ACR core set. This index was calculated as minimum of either a) % change in TJC, b) % change in SJC, or c) the median % change of remaining 5 ACR core criteria: If ≥3 components of the 5 ACR core criteria were missing, then c) was set to missing; if any of 3 components a), b), or c) were missing, then ACR-N was set to missing. Percentage of improvement was truncated to range of -100 to 100 to minimize impact of outliers (greater values indicate greater % improvement) and negative scores indicate a decline. Least Squares (LS) means were calculated using analysis of covariance (ANCOVA) with treatment and region as fixed factors and baseline Disease Activity Score based on 28 joint counts -CRP (DAS28-CRP) as a covariate.
Time Frame: Baseline through Week 24
Population: All randomized participants with evaluable ACR-N data. Modified Baseline Observation Carried Forward (mBOCF) was used to impute missing post-baseline values. Data after Week 16 for Week 16 NR were not included.
Measure: Least Squares Mean (Standard Error); unit: percentage of improvement
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 153 | 146 | 153
percentage of improvement | -9.03 (4.00) | -8.03 (4.11) | -12.72 (4.00)

4. Secondary Outcome: Change From Baseline to Week 24 in Tender Joint Count (68 Joint Count)
Description: Tender joint count is the number of tender and painful joints determined for each participant by examination of 68 joints. Joints were assessed by pressure and joint manipulation on physical examination. Participants were asked for pain sensations on these manipulations and watched for spontaneous pain reactions. Any positive response on pressure, movement, or both was translated into a single tender-versus-nontender dichotomy. LS means were calculated using ANCOVA with treatment and region as fixed factors and baseline as a covariate.
Time Frame: Baseline, Week 24
Population: All randomized participants with evaluable tender joint count data. mBOCF was used to impute missing post-baseline values. Data after Week 16 for Week 16 NR were not included.
Measure: Least Squares Mean (Standard Error); unit: joint counts
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 153 | 147 | 154
joint counts | -6.37 (1.40) | -6.08 (1.42) | -6.56 (1.38)

5. Secondary Outcome: Change From Baseline to Week 24 in Swollen Joint Count (66 Joint Count)
Description: Swollen joint count is the number of swollen joints determined for each participant by examination of 66 joints. Joints were classified as either swollen or not swollen. Swelling was defined as palpable fluctuating synovitis of the joint. LS means were calculated using ANCOVA with treatment and region as fixed factors and baseline as a covariate.
Time Frame: Baseline, Week 24
Population: All randomized participants with evaluable swollen joint count data. mBOCF was used to impute missing post-baseline values. Data after Week 16 for Week 16 NR were not included.
Measure: Least Squares Mean (Standard Error); unit: joint counts
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 153 | 147 | 154
joint counts | -6.02 (0.98) | -5.64 (1.00) | -5.41 (0.98)

6. Secondary Outcome: Change From Baseline to Week 24 in Participant's Assessment of Pain [Visual Analog Scale (VAS)]
Description: Participant's assessment of their current arthritis pain using VAS ranged from 0 millimeters (mm) (no pain) to 100 mm (worst possible pain). A decrease in pain score indicated an improvement in the participant's condition. LS means were calculated using ANCOVA with treatment and region as fixed factors and baseline as a covariate.
Time Frame: Baseline, Week 24
Population: All randomized participants with evaluable participant's assessment of pain data. mBOCF was used to impute missing post-baseline values. Data after Week 16 for Week 16 NR were not included.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 153 | 146 | 153
mm | -9.89 (2.10) | -9.15 (2.15) | -5.76 (2.10)

7. Secondary Outcome: Change From Baseline to Week 24 in Participant's Global Assessment of Disease Activity (VAS)
Description: Participant's assessment of their current arthritis disease activity using VAS ranged from 0 mm (no arthritis activity) to 100 mm (extremely active arthritis). A decrease in disease activity score indicated an improvement in the participant's condition. LS means were calculated using ANCOVA with treatment and region as fixed factors and baseline as a covariate.
Time Frame: Baseline, Week 24
Population: All randomized participants with evaluable participant's global assessment of disease activity data. mBOCF was used to impute missing post-baseline values. Data after Week 16 for Week 16 NR were not included.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 153 | 146 | 153
mm | -11.29 (2.14) | -8.72 (2.19) | -7.12 (2.13)

8. Secondary Outcome: Change From Baseline to Week 24 in Physician's Global Assessment of Disease Activity (VAS)
Description: Physician's assessment of the participant's current arthritis disease activity using VAS ranged from 0 mm (no arthritis activity) to 100 mm (extremely active arthritis). A decrease in disease activity score indicated an improvement in the participant's condition. LS means were calculated using ANCOVA with treatment and region as fixed factors and baseline as a covariate.
Time Frame: Baseline, Week 24
Population: All randomized participants with evaluable physician's global assessment of disease activity data. mBOCF was used to impute missing post-baseline values. Data after Week 16 for Week 16 NR were not included.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 147 | 140 | 150
mm | -15.90 (2.16) | -16.38 (2.23) | -13.17 (2.13)

9. Secondary Outcome: Change From Baseline to Week 24 in Health Assessment Questionnaire-Disability Index (HAQ-DI)
Description: The HAQ-DI questionnaire assesses the participant's self-perception on the degree of difficulty [0 (without any difficulty), 1 (with some difficulty), 2 (with much difficulty), and 3 (unable to do)] when dressing and grooming, arising, eating, walking, hygiene, reaching, gripping, and performing other daily activities. Scores for each functional area were averaged to calculate HAQ-DI scores, which ranged from 0 (no disability) to 3 (severe disability). A decrease in HAQ-DI score indicated an improvement in the participant's condition. LS means were calculated using ANCOVA with treatment and region as fixed factors and baseline as a covariate.
Time Frame: Baseline, Week 24
Population: All randomized participants with evaluable HAQ-DI data. mBOCF was used to impute missing post-baseline values. Data after Week 16 for Week 16 NR were not included.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 153 | 146 | 153
units on a scale | -0.13 (0.05) | -0.09 (0.05) | -0.08 (0.05)

10. Secondary Outcome: Change From Baseline to Week 24 in Disease Activity Score Based on 28 Joint Count and C-Reactive Protein Level (DAS28-CRP)
Description: Disease Activity Score (DAS) modified to include 28 joint count (DAS28) consisted of composite score of following variables: tender joint count (TJC28), swollen joint count (SJC28), CRP (milligrams per liter), and participant's global assessment of disease activity using VAS (participant global VAS). DAS28-CRP=0.56*square root (sqrt)(TJC28)+0.28*sqrt(SJC28)+0.36*natural log(CRP+1)+0.014*participant global VAS+0.96. Scores ranged from 1.0 to 9.4, where lower scores indicated less disease activity and remission is DAS28-CRP <2.6. A decrease in DAS28-CRP indicated an improvement in participant's condition. LS means were calculated using ANCOVA with treatment and region as fixed factors and baseline as a covariate.
Time Frame: Baseline, Week 24
Population: All randomized participants with evaluable DAS28-CRP data. mBOCF was used to impute missing post-baseline values. Data after Week 16 for Week 16 NR were not included.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 152 | 146 | 152
units on a scale | -0.76 (0.12) | -0.79 (0.13) | -0.72 (0.12)

11. Secondary Outcome: Percentage of Participants With DAS28-CRP Based European League Against Rheumatism (EULAR) Response
Description: EULAR Responder index categorizes clinical response based on improvement since baseline in DAS28-CRP. DAS28-CRP=0.56*sqrt(TJC28)+0.28*sqrt(SJC28)+0.36*natural log(CRP+1)+0.014*participant global VAS+0.96. DAS28-CRP scores range from 1.0-9.4, where lower scores indicated less disease activity. High disease activity: DAS28-CRP >5.1, low disease activity: DAS28-CRP <3.2, and remission: DAS28-CRP <2.6. Participants are categorized as EULAR responders or NR based on improvement of DAS28-CRP scores from baseline. EULAR DAS28-CRP responder index defines a good (absolute: <3.2 or >1.2 improvement from baseline), moderate (absolute: 3.2-5.1 or 0.6-1.2 improvement from baseline), or no response (absolute: >5.1 or <0.6 improvement from baseline). Percentage of participants with DAS28-CRP based EULAR response = ( number of participants with specific response) / (number of participants analyzed in the group) * 100.
Time Frame: Baseline through Week 24
Population: All randomized participants with evaluable EULAR response data. Modified Last Observation Carried Forward (mLOCF) was used to impute missing post-baseline values. Data after Week 16 for Week 16 NR were not included.
Measure: Number; unit: percentage of participants
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 152 | 146 | 152
percentage of participants
  Good | 11.8 | 9.6 | 8.6
  Moderate | 36.2 | 36.3 | 36.2
  No response | 52.0 | 54.1 | 55.3

12. Secondary Outcome: Change From Baseline to Week 24 in Medical Outcomes Study 36-Item Short Form (SF-36) Health Survey Domain and Summary Scores
Description: SF-36 is a health-related survey that assesses participant's quality of life and consists of 36 questions covering 8 health domains: physical functioning, bodily pain, role limitations due to physical problems and emotional problems, general health, mental health, social functioning, vitality, 2 component scores (CS), physical CS (PCS) and mental CS (MCS). Domain scores calculated by summing each item for each domain and transforming scores into 0-100 scale; higher scores indicated better health status. If < 50% of the questions within a domain were answered, the raw score were not calculated. PCS score consisted of physical functioning, bodily pain, role-physical, and general health scales. MCS score consisted of social functioning, vitality, mental health, and role-emotional scales. Both PCS and MCS range from 0-100 with higher score indicating better mental or physical health. LS means were calculated using ANCOVA with treatment, region as fixed factors and baseline as a covariate.
Time Frame: Baseline, Week 24
Population: All randomized participants with evaluable SF-36 domain and summary scores. mBOCF was used to impute missing post-baseline values. Data after Week 16 for Week 16 NR were not included.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 146 | 138 | 149
units on a scale
  Physical Functioning | 1.81 (0.78) | 1.78 (0.82) | 1.00 (0.77)
  Bodily Pain | 2.36 (0.75) | 2.95 (0.78) | 1.97 (0.74)
  Role Limitations due to Physical Problems | 1.92 (0.72) | 2.08 (0.75) | 0.35 (0.72)
  Role Limitations due to Emotional Problems | 1.07 (0.97) | 2.55 (1.01) | 1.19 (0.96)
  General Health Perception | 1.90 (0.64) | 0.91 (0.67) | 1.88 (0.64)
  Mental Health | 0.83 (0.85) | 1.57 (0.88) | 0.98 (0.84)
  Social Function | 2.51 (0.87) | 1.68 (0.91) | 1.32 (0.86)
  Vitality | 2.71 (0.77) | 2.40 (0.80) | 2.05 (0.76)
  PCS | 2.30 (0.71) | 1.83 (0.74) | 1.21 (0.71)
  MCS | 1.22 (0.87) | 1.86 (0.90) | 1.38 (0.86)

13. Secondary Outcome: Change From Baseline to Week 24 in Brief Fatigue Inventory (BFI) Individual Items and Impact Scores
Description: The BFI is a brief participant-reported questionnaire for the rapid assessment of fatigue severity and the impact of fatigue on daily functioning in the past 24 hours. The BFI contains 10 items; however, the first item is not included in the scoring of the scale as it asks about usual fatigue over the past week with the participant answering 'yes' or 'no'. The remaining 9 items assess fatigue severity (3 items) and impact of fatigue on daily functioning (6 items) using an 11-point numeric scale, with 0 = no fatigue and 10 = fatigue as bad as you can imagine. The fatigue impact subscale score is the average of the non-missing responses to 6 items: general activity, mood, walking ability, normal work, relations with other people, and enjoyment of life. If more than 3 items within the fatigue impact subscale were not answered by a participant, the subscale is set to missing. LS means were calculated using ANCOVA with treatment and region as fixed factors and baseline as a covariate.
Time Frame: Baseline, Week 24
Population: All randomized participants with evaluable BFI data. mBOCF was used to impute missing post-baseline values. Data after Week 16 for Week 16 NR were not included.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 146 | 138 | 149
units on a scale
  Fatigue - Now | -0.68 (0.12) | -0.55 (0.12) | -0.60 (0.12)
  Fatigue - Usual | -0.65 (0.11) | -0.58 (0.11) | -0.56 (0.11)
  Fatigue - Worst | -0.75 (0.12) | -0.65 (0.12) | -0.72 (0.12)
  General Activity | -0.55 (0.12) | -0.50 (0.12) | -0.52 (0.12)
  Mood | -0.54 (0.12) | -0.35 (0.12) | -0.35 (0.12)
  Walking Ability | -0.53 (0.12) | -0.38 (0.13) | -0.36 (0.12)
  Normal Work | -0.60 (0.12) | -0.46 (0.12) | -0.42 (0.12)
  Relations with Other People | -0.41 (0.12) | -0.43 (0.12) | -0.29 (0.12)
  Enjoyment of Life | -0.53 (0.13) | -0.55 (0.13) | -0.41 (0.13)
  Fatigue Impact Subscale | -0.52 (0.11) | -0.43 (0.11) | -0.39 (0.11)

14. Secondary Outcome: Change From Baseline to Week 24 in Brief Pain Inventory Short Form (BPI-SF) Individual Items and Interference Scores
Description: The BPI-SF is a self-reported scale that measures the severity of pain based on the worst pain, least pain, average pain experienced during the past 24 hours and pain based on the pain right now, with scores ranging from 0 (no pain) to 10 (pain as severe as you can imagine). Pain interference score is the average of the responses in the past 24 hours to 7 items: general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life [each item scored from 0 (does not interfere) to 10 (completely interferes)]. If more than 3 items of the Pain Interference Score are not answered by a participant, the score is set to missing. LS means were calculated using ANCOVA with treatment and region as fixed factors and baseline as a covariate.
Time Frame: Baseline, Week 24
Population: All randomized participants with evaluable BPI-SF scores. mBOCF was used to impute missing post-baseline values. Data after Week 16 for Week 16 NR were not included.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 146 | 138 | 149
units on a scale
  Pain - Worst | -0.9 (0.2) | -0.8 (0.2) | -0.4 (0.2)
  Pain - Least | -0.5 (0.2) | -0.5 (0.2) | -0.1 (0.2)
  Pain - Average | -0.7 (0.2) | -0.7 (0.2) | -0.3 (0.2)
  Pain - Now: number analyzed (Participants) | 146 | 137 | 149
  Pain - Now | -0.8 (0.2) | -0.5 (0.2) | -0.3 (0.2)
  General Activity: number analyzed (Participants) | 146 | 137 | 149
  General Activity | -0.7 (0.2) | -0.4 (0.2) | -0.3 (0.2)
  Mood: number analyzed (Participants) | 146 | 137 | 149
  Mood | -0.6 (0.2) | -0.2 (0.2) | -0.0 (0.2)
  Walking Ability: number analyzed (Participants) | 146 | 137 | 149
  Walking Ability | -0.8 (0.2) | -0.4 (0.2) | -0.4 (0.2)
  Normal Work: number analyzed (Participants) | 146 | 137 | 149
  Normal Work | -0.7 (0.2) | -0.4 (0.2) | -0.2 (0.2)
  Relations with Other People: number analyzed (Participants) | 146 | 137 | 149
  Relations with Other People | -0.3 (0.2) | -0.2 (0.2) | -0.1 (0.2)
  Sleep: number analyzed (Participants) | 146 | 137 | 149
  Sleep | -0.7 (0.2) | -0.3 (0.2) | -0.4 (0.2)
  Enjoyment of Life: number analyzed (Participants) | 146 | 137 | 149
  Enjoyment of Life | -0.7 (0.2) | -0.4 (0.2) | -0.4 (0.2)
  Pain Interference Score: number analyzed (Participants) | 146 | 137 | 149
  Pain Interference Score | -0.6 (0.2) | -0.3 (0.2) | -0.3 (0.2)

15. Secondary Outcome: Change From Baseline to Week 24 in Duration of Morning Stiffness (Minutes)
Description: The Investigator asks participants about the duration of their morning stiffness (in minutes) in and around the joints and records the duration. The Investigator should ask participants about duration of morning stiffness on the day prior to the study visit to capture actual symptoms. If morning stiffness duration is longer than 12 hours (720 minutes), it was truncated to 720 minutes for statistical presentations and analyses.LS means were calculated using ANCOVA with treatment and region as fixed factors and baseline as a covariate.
Time Frame: Baseline, Week 24
Population: All randomized participants with evaluable morning stiffness data; mBOCF was used to impute missing post-baseline values. Data after Week 16 for Week 16 NR were not included.
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 141 | 138 | 139
minutes | -20.6 (11.5) | -1.0 (11.7) | -18.0 (11.9)

16. Secondary Outcome: Time to ACR20 Response
Time Frame: Baseline through Week 24
Population: Zero participants analyzed. Time to ACR20 data not collected for analysis.
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 0 | 0 | 0

17. Secondary Outcome: Change From Baseline to Week 24 in Absolute B Cell Counts
Description: Cell-surface marker cluster designation (CD) 3 negative, CD20 positive (CD3-CD20+) defines total mature B cells. B-lymphocyte antigen CD20 is an activated-glycosylated phosphoprotein expressed on the surface of all mature B cells. Baseline B cell count is the average of the values on or prior to the date of first injection of study treatment, including unscheduled visits. A positive or negative change indicated an increase or decrease, respectively in B cell count. LS means were calculated using ANCOVA with treatment and region as fixed factors and baseline as a covariate.
Time Frame: Baseline, Week 24
Population: All randomized participants with evaluable CD3-CD20+ B cell counts. mLOCF was used to impute missing post-baseline values. Data after Week 16 for Week 16 NR were not included.
Measure: Least Squares Mean (Standard Error); unit: cells/microliter (cells/µL)
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 151 | 147 | 154
cells/microliter (cells/µL) | -55.3 (9.9) | -65.8 (10.1) | 3.2 (9.8)

18. Secondary Outcome: Change From Baseline to Week 24 in Serum Immunoglobulin (Ig) Levels
Description: Immunoglobulin (Ig), or antibodies, are large proteins used by the immune system to identify and neutralize foreign particles such as bacteria and viruses. Their normal blood levels indicate proper immune status. Change from baseline in serum immunoglobulin A (IgA), immunoglobulin G (IgG), and immunoglobulin M (IgM) levels are reported. A negative change indicated a decrease in Ig levels. LS means were calculated using ANCOVA with treatment and region as fixed factors and baseline as a covariate.
Time Frame: Baseline, Week 24
Population: All randomized participants with evaluable serum Ig data. mLOCF was used to impute missing post-baseline values. Data after Week 16 for Week 16 NR were not included.
Measure: Least Squares Mean (Standard Error); unit: grams/liter (g/L)
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 151 | 146 | 153
grams/liter (g/L)
  IgA | -0.330 (0.049) | -0.324 (0.050) | 0.003 (0.049)
  IgG | -0.955 (0.161) | -0.978 (0.163) | 0.058 (0.158)
  IgM | -0.273 (0.043) | -0.239 (0.044) | -0.019 (0.042)

19. Secondary Outcome: Population Pharmacokinetics (PK): Constant Clearance
Description: Population estimate of constant clearance as determined by population PK analysis. A 2-compartment model was used in PK modeling. Constant clearance is the PK parameter which describes the linear elimination of LY2127399 from serum.
Time Frame: Baseline through Week 24
Population: All randomized participants who received at least 1 dose of LY2127399 with evaluable LY2127399 PK data.
Measure: Mean (Standard Error); unit: milliliters/hour (mL/h)
Groups:
- 120 mg LY2127399: A loading dose of 240 mg (2 injections of 120 mg) of LY2127399 followed by maintenance dosing of 120 mg of LY2127399 administered SC Q4W for 24 weeks or a loading dose of 180 mg of LY2127399 (2 injections of 90 mg) followed by maintenance dosing of 90 mg of LY2127399 administered SC Q2W for 24 weeks. At Week 16, responders received 1 injection of 120 mg of LY2127399 and 1 injection of placebo, followed by 120 mg of LY2127399 Q4W for the rest of the 24-week treatment period or 1 injection of 90 mg of LY2127399 and 1 injection of placebo, followed by 90 mg of LY2127399 Q2W for the rest of the 24-week treatment period.
  At Week 16, NR received 1 injection of 90 mg of LY2127399 and 1 injection of placebo, followed by 90 mg of LY2127399 Q2W for the rest of the 24-week treatment period.
Arm/Group | 120 mg LY2127399
Number analyzed (Participants) | 309
milliliters/hour (mL/h) | 4.16 (3.58) [3.44 to 3.78]

20. Secondary Outcome: Percentage of Participants Developing Anti-LY2127399 Antibodies
Description: Participants with treatment-emergent anti-drug antibody (ADA) were participants who had any sample from baseline up to and through Week 52 that was a 4-fold increase (2-dilution increase) in immunogenicity titer over baseline titer, or participants who tested negative at baseline and positive post-baseline (at titer of ≥1:20). Percentage of participants with ADA = (number of participants with treatment-emergent ADA) / (number of participants assessed) * 100.
Time Frame: Baseline through Week 24
Population: All randomized participants who received at least 1 dose of study drug with an evaluable baseline ADA result and a post-baseline ADA result. Participants missing an evaluable baseline result with all negative post-baseline results were included. Data after Week 16 for Week 16 NR were not included.
Measure: Number; unit: percentage of participants
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 153 | 147 | 154
percentage of participants | 3.9 | 4.8 | 3.9

21. Secondary Outcome: Change From Baseline to Week 24 in CRP
Description: CRP is an indicator of inflammation. A negative change indicated an improvement in the participant's condition. LS means were calculated using ANCOVA with treatment and region as fixed factors and baseline as a covariate.
Time Frame: Baseline, Week 24
Population: All randomized participants with evaluable CRP data. mBOCF was used to impute missing post-baseline values. Data after Week 16 for Week 16 NR were not included.
Measure: Least Squares Mean (Standard Error); unit: milligrams/liter (mg/L)
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 152 | 147 | 154
milligrams/liter (mg/L) | 2.91 (1.83) | 0.95 (1.87) | 2.93 (1.81)

ADVERSE EVENTS:
Groups:
- LY 120 mg Q4W, Randomized Treatment Period: A loading dose of 240 mg of LY2127399 (2 injections of 120 mg) followed by maintenance dosing of 120 mg of LY2127399 administered SC Q4W for 24 weeks. At Week 16, responders received 1 injection of 120 mg of LY2127399 and 1 injection of placebo, followed by 120 mg of LY2127399 Q4W for the rest of the 24-week treatment period. For blinding purposes, participants alternated injections of LY2127399 and injections of placebo Q2W.
  The Randomized Treatment Period was defined as the time all data was collected during the treatment period, excluding the data collected after the date of the Week 16 injection for the Week 16 NR.
- LY 90 mg Q2W, Randomized Treatment Period: A loading dose of 180 mg of LY2127399 (2 injections of 90 mg) followed by maintenance dosing of 90 mg of LY2127399 administered SC Q2W for 24 weeks. At Week 16, responders received 1 injection of 90 mg of LY2127399 and 1 injection of placebo, followed by 90 mg of LY2127399 Q2W for the rest of the 24-week treatment period.
  The Randomized Treatment Period was defined as the time all data was collected during the treatment period, excluding the data collected after the date of the Week 16 injection for the Week 16 NR.
- Placebo, Randomized Treatment Period: A loading dose of 2 injections of placebo followed by maintenance dosing of 1 injection of placebo administered SC Q2W for 24 weeks. At Week 16, responders received 2 injections of placebo, followed by 1 injection of placebo Q2W for the rest of the 24-week treatment period.
  The Randomized Treatment Period was defined as the time all data was collected during the treatment period, excluding the data collected after the date of the Week 16 injection for the Week 16 NR.
- LY 120 mg Q4W, Rescue Period: A loading dose of 240 mg of LY2127399 (2 injections of 120 mg) followed by maintenance dosing of 120 mg of LY2127399 administered SC Q4W for 16 weeks. For blinding purposes, participants alternated injections of LY2127399 and injections of placebo Q2W.
  At Week 16, NR received 1 injection of 90 mg of LY2127399 and 1 injection of placebo, followed by 90 mg of LY2127399 Q2W for the rest of the 24-week treatment period.
  The Rescue Treatment Period was defined as all data collected after the date of the Week 16 injection during the treatment period for Week 16 NR.
- LY 90 mg Q2W, Rescue Period: A loading dose of 180 mg of LY2127399 (2 injections of 90 mg) followed by maintenance dosing of 90 mg of LY2127399 administered SC Q2W for 16 weeks.
  At Week 16, NR received 1 injection of 90 mg of LY2127399 and 1 injection of placebo, followed by 90 mg of LY2127399 Q2W for the rest of the 24-week treatment period.
  The Rescue Treatment Period was defined as all data collected after the date of the Week 16 injection during the treatment period for Week 16 NR.
- Placebo, Rescue Period: A loading dose of 2 injections of placebo followed by maintenance dosing of 1 injection of placebo administered SC Q2W for 16 weeks.
  At Week 16, NR received a loading dose of 180 mg of LY2127399 (2 injections of 90 mg), followed by 90 mg of LY2127399 Q2W for the rest of the 24-week treatment period.
  The Rescue Treatment Period was defined as all data collected after the date of the Week 16 injection during the treatment period for Week 16 NR.
- LY 120 mg Q4W, Follow-up Period: A loading dose of 240 mg (2 injections of 120 mg) of LY2127399 followed by maintenance dosing of 120 mg of LY2127399 administered SC Q4W for 24 weeks. At Week 16, responders received 1 injection of 120 mg of LY2127399 and 1 injection of placebo, followed by 120 mg of LY2127399 Q4W for the rest of the 24-week treatment period. For blinding purposes, participants alternated injections of LY2127399 and injections of placebo Q2W.
  The Post-Treatment Follow-Up Period started after Week 24 or the early discontinuation visit and lasted up to 48 weeks following the last injection of study treatment.
- LY 90 mg Q2W, Follow-up Period: A loading dose of 180 mg of LY2127399 (2 injections of 90 mg) followed by maintenance dosing of 90 mg of LY2127399 administered SC Q2W for 24 weeks. At Week 16, both responders and NR received 1 injection of 90 mg of LY2127399 and 1 injection of placebo, followed by 90 mg of LY2127399 Q2W for the rest of the 24-week treatment period.
  The Post-Treatment Follow-Up Period started after Week 24 or the early discontinuation visit and lasted up to 48 weeks following the last injection of study treatment.
- Placebo, Follow-up Period: A loading dose of 2 injections of placebo followed by maintenance dosing of 1 injection of placebo administered SC Q2W for 24 weeks. At Week 16, responders received 2 injections of placebo, followed by 1 injection of placebo Q2W for the rest of the 24-week treatment period.
  The Post-Treatment Follow-Up Period started after Week 24 or the early discontinuation visit and lasted up to 48 weeks following the last injection of study treatment.
- LY 120 mg Q4W to LY 90 mg Q2W (Week 16), Follow-up Period: A loading dose of 240 mg of LY2127399 (2 injections of 120 mg) followed by maintenance dosing of 120 mg of LY2127399 administered SC Q4W for 16 weeks. For blinding purposes, participants alternated injections of LY2127399 and injections of placebo Q2W.
  At Week 16, NR received 1 injection of 90 mg of LY2127399 and 1 injection of placebo, followed by 90 mg of LY2127399 Q2W for the rest of the 24-week treatment period.
  The Post-Treatment Follow-Up Period started after Week 24 or the early discontinuation visit and lasted up to 48 weeks following the last injection of study treatment.
- Placebo to LY 90 mg Q2W (Week 16), Follow-up Period: A loading dose of 2 injections of placebo followed by maintenance dosing of 1 injection of placebo administered SC Q2W for 16 weeks.
  At Week 16, NR received a loading dose of 180 mg of LY2127399 (2 injections of 90 mg), followed by 90 mg of LY2127399 Q2W for the rest of the 24-week treatment period.
  The Post-Treatment Follow-Up Period started after Week 24 or the early discontinuation visit and lasted up to 48 weeks following the last injection of study treatment.
Arm/Group | LY 120 mg Q4W, Randomized Treatment Period | LY 90 mg Q2W, Randomized Treatment Period | Placebo, Randomized Treatment Period | LY 120 mg Q4W, Rescue Period | LY 90 mg Q2W, Rescue Period | Placebo, Rescue Period | LY 120 mg Q4W, Follow-up Period | LY 90 mg Q2W, Follow-up Period | Placebo, Follow-up Period | LY 120 mg Q4W to LY 90 mg Q2W (Week 16), Follow-up Period | Placebo to LY 90 mg Q2W (Week 16), Follow-up Period
Serious Adverse Events (participants affected / at risk) | 7/153 | 6/147 | 6/154 | 1/23 | 2/33 | 1/37 | 1/43 | 1/36 | 3/44 | 0/3 | 0/7
Other Adverse Events (participants affected / at risk) | 71/153 | 51/147 | 61/154 | 10/23 | 11/33 | 16/37 | 6/43 | 11/36 | 14/44 | 0/3 | 1/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY 120 mg Q4W, Randomized Treatment Period (N=153) | LY 90 mg Q2W, Randomized Treatment Period (N=147) | Placebo, Randomized Treatment Period (N=154) | LY 120 mg Q4W, Rescue Period (N=23) | LY 90 mg Q2W, Rescue Period (N=33) | Placebo, Rescue Period (N=37) | LY 120 mg Q4W, Follow-up Period (N=43) | LY 90 mg Q2W, Follow-up Period (N=36) | Placebo, Follow-up Period (N=44) | LY 120 mg Q4W to LY 90 mg Q2W (Week 16), Follow-up Period (N=3) | Placebo to LY 90 mg Q2W (Week 16), Follow-up Period (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyomyositis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somatoform disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LY 120 mg Q4W, Randomized Treatment Period (N=153) | LY 90 mg Q2W, Randomized Treatment Period (N=147) | Placebo, Randomized Treatment Period (N=154) | LY 120 mg Q4W, Rescue Period (N=23) | LY 90 mg Q2W, Rescue Period (N=33) | Placebo, Rescue Period (N=37) | LY 120 mg Q4W, Follow-up Period (N=43) | LY 90 mg Q2W, Follow-up Period (N=36) | Placebo, Follow-up Period (N=44) | LY 120 mg Q4W to LY 90 mg Q2W (Week 16), Follow-up Period (N=3) | Placebo to LY 90 mg Q2W (Week 16), Follow-up Period (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (6) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 1 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 2 (6) | 5 (18) | 4 (21) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 4 (6) | 7 (19) | 0 (0) | 0 (0) | 0 (0) | 3 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 4 (4) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenoiditis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alveolar osteitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 3 (3) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 5 (6) | 2 (2) | 7 (7) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 9 (10) | 7 (7) | 9 (11) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 5 (5) | 6 (6) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitamin d deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 8 (9) | 7 (7) | 11 (13) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/29 (1) | 0/22 (0) | 0/24 (0) | 0/4 (0) | 0/5 (0) | 0/4 (0) | 0/11 (0) | 0/8 (0) | 0/10 (0) | 0/0 (0) | 0/0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 7 (8) | 2 (2) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 0/124 (0) | 0/125 (0) | 0/130 (0) | 1/19 (1) | 0/28 (0) | 0/33 (0) | 0/32 (0) | 0/28 (0) | 0/34 (0) | 0 (0) | 0 (0)
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
This study has been terminated not based on safety concerns, but due to insufficient efficacy. Early termination led to lower than expected enrollment and was responsible for the large number of discontinuation reason as Sponsor Decision.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days